CLINICAL TRIAL: NCT01231646
Title: Does Valproate Increase Levels of Folate Receptor Autoantibodies in Women?
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Epilepsy Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 10-266A
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Epilepsy; Psychiatric or Mood Diseases or Conditions
Keywords: Folate Receptor Autoantibodies; Epilepsy; Psychiatric conditions
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lamotrigine: No intervention
  Interventions: Other: No intervention
- Valproate: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. This is a cross-sectional study.

SUMMARY:
Women who take folate (folic acid) before getting pregnant can lower the risk of giving birth to infant with certain birth defects. However, some medications may affect the action of folate. The purpose of this study is to compare the effect of two anti-epileptic drugs on how folate works in our body.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-50 years inclusive who are taking valproate or lamotrigine for neurologic or psychiatric conditions
* Valproate of lamotrigine must be used as monotherapy at stable doses for 6 weeks prior to the study for the neurologic or psychiatric illness; medications taken for other reasons are not excluded.

Exclusion Criteria:

* Women with prior exposure to valproate or lamotrigine if they are taking lamotrigine or valproate respectively.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients in epilepsy and/or psychiatric clinics
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Harden, MD, Principal Investigator — North Shore-Long Island Jewish Medical Center
Locations (1):
- North Shore Long Island Jewish Health System, Great Neck, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine: Women on lamotrigine monotherapy or polytherapy, and had never been exposed to valproate.
- Valproate: Women on valproate monotherapy or polytherapy, and had never been exposed to lamotrigine.
Period: Overall Study
Arm/Group | Lamotrigine | Valproate
Started | 28 | 10
Completed | 28 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Valproate | Total
Number analyzed (Participants) | 28 | 10 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10.22) | 39.1 (7.77) | 34.7 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 10 | 38
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.95 (4.3) | 30.47 (7.2) | 26.44 (5.77)

OUTCOME MEASURES:

1. Primary Outcome: Levels of Folate Receptor Autoantibodies
Description: ELISA assays using immobilized folate receptor protein were performed to determine the titers of immunoglobulin G, immunoglobulin M, and combined immunoglobulin G and immunoglobulin M to folate receptor in serum samples collected from both groups of women.
Time Frame: On the same day after informed consent was obtained
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Lamotrigine | Valproate
Number analyzed (Participants) | 27 | 10
ug/mL
  Immunoglobulin G | 35.33 (27.14) | 35.21 (20.57)
  Immunoglobulin M | 44.3 (34.18) | 41.81 (33.13)
  Immunoglobulin G and Immunoglobulin M | 79.62 (50.12) | 77.06 (46.00)

ADVERSE EVENTS:
Description: This is a cross-sectional 1 visit study. No Adverse Event were collected or assessed.
Arm/Group | Lamotrigine | Valproate
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No